CLINICAL TRIAL: NCT04145609
Title: Strategies to Stop Acute Kidney Injury (AKI)-Acute Kidney Disease (AKD) -Chronic Kidney Disease (CKD) Continuum - Policy The Intensified AKD Care to Reduce CKD
Brief Title: Intensified Acute Kidney Disease Care to Reduce Chronic Kidney Disease
Acronym: ISACC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other); Taipei Medical University (Other)
Responsible Party: Principal Investigator, Shuang-Ho Hospital, the EIRAP project, Stop AKI-AKD-CKD continuum in Taiwan: from precision medicine to policy decision (EIRAP study), Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: N201905047
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Acute Kidney Injury; Renal Insufficiency, Chronic; Acute Kidney Disease; Decision Support Systems, Clinical
Keywords: Acute Kidney Injury; Acute Kidney Disease; Chronic Kidney Disease; AKI; AKD; CKD; Decision Support Systems, Clinical; CDS
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency, Chronic | interventions — Ambulatory Care Facilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensified care (Experimental): Experimental: Multidisciplinary team (MDT) care + Acute kidney disease (AKD) clinic Participants randomized to this arm will receive multidisciplinary team (MDT) care by a specialized medical team which is composed of nephrologist, pharmacist and dietitian. Besides intensified care, participants of this arm receive evaluation of biochemical and physiological renal function more frequently. In order to provide seamless care of this group, post-discharge acute kidney disease (AKD) clinic will also be arranged for them. Clinic visits consist of evaluation of renal function, reconciliation of medication and steering necessity of renal replacement therapy.
  Interventions: Behavioral: Multidisciplinary team (MDT) care and Acute kidney disease (AKD) clinic
- Usual care (No Intervention): No intervention: Usual care Participants randomized to this arm will receive usual care according to the medical decisions of principal care physician. Nephrologist consultation and nephrology outpatient clinic follow-up will be allowed. However, this group of patient will not have access to MDT care and AKD clinic.

INTERVENTIONS:
Behavioral: Multidisciplinary team (MDT) care and Acute kidney disease (AKD) clinic — Multidisciplinary team (MDT) care: NPDS care model Acute kidney disease (AKD) clinic: layered approach
  Arms: Intensified care

SUMMARY:
Strategies to stop AKI-AKD-CKD continuum - Policy is one of the collaborative projects, Strategies to stop AKI-AKD-CKD continuum, Epidemiology, Immunology, Repair, Artificial intelligence, and Policy (EIRAP). It is aimed to study effective interventional strategies that lower the incidence of CKD among patients with AKD. The intensified AKD care to reduce CKD (ISACC trial) is a prospective, open-labeled, randomized controlled trial is designed to evaluate the efficacy of multidisciplinary team care (MDT) model and acute kidney disease (AKD) clinic visits

DETAILED DESCRIPTION:
Acute kidney disease (AKD), defined as the ongoing renal function impairment between 7 days and 90 days following AKI, has been proposed as a window of intervention to prevent the occurrence of CKD. However, the effective therapeutic strategies of AKD care remain to be developed. We intend to conduct a prospective, randomized, open-label, behavioral interventional trial to validate the efficacy of multidisciplinary team (MDT) care model which aims to improve AKD care and to reduce de novo CKD incidence.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 yrs
* Severe AKD: Stage 2, Stage 3 and Dialysis-requiring AKD (AKD-D)

Exclusion Criteria:

* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Major adverse kidney event | 90days
  Proportion of MAKE
  * Renal progression to CKD
  * Chronic dialysis (any 1 outpatient dialysis after discharge)
  * Death

SECONDARY OUTCOMES:
Mortality | 30days, 60days, 90days, 180days, 360 days, 3years
  Proportion of death
Chronic dialysis | 90days, 180days, 360 days, 3years
  Proportion of chronic dialysis
Renal progression | 90days, 180days, 360 days, 3years
  Proportion of renal progression to CKD
Time to MAKE | 90days, 180days, 1year (360days)
  Time to MAKE
Time to death | 90days, 180days, 1year (360days)
  Time to death
Time to chronic dialysis | 90days, 180days, 1year (360days)
  Time to chronic dialysis
Time to renal progression to CKD | 90days, 180days, 1year (360days)
  Time to renal progression to CKD
Time to first ER visit | 90days, 180days, 1year (360days)
  Time to first ER visit
Time to first rehospitalization | 90days, 180days, 1year (360days)
  Time to first rehospitalization
Time to first recurrence of AKI | 90days, 180days, 1year (360days)
  Time to first recurrence of AKI
Proportion of MACE | 30days, 60days, 90days, 180days, 360 days, 3years
  CVA, AMI, CHF, or cardiac revascularization procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Szu Wu, Study Chair — Shuang Ho Hospital, Taipei Medical University

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Chawla LS, Bellomo R, Bihorac A, Goldstein SL, Siew ED, Bagshaw SM, Bittleman D, Cruz D, Endre Z, Fitzgerald RL, Forni L, Kane-Gill SL, Hoste E, Koyner J, Liu KD, Macedo E, Mehta R, Murray P, Nadim M, Ostermann M, Palevsky PM, Pannu N, Rosner M, Wald R, Zarbock A, Ronco C, Kellum JA; Acute Disease Quality Initiative Workgroup 16.. Acute kidney disease and renal recovery: consensus report of the Acute Disease Quality Initiative (ADQI) 16 Workgroup. Nat Rev Nephrol. 2017 Apr;13(4):241-257. doi: 10.1038/nrneph.2017.2. Epub 2017 Feb 27. PMID 28239173
- [Background] See EJ, Jayasinghe K, Glassford N, Bailey M, Johnson DW, Polkinghorne KR, Toussaint ND, Bellomo R. Long-term risk of adverse outcomes after acute kidney injury: a systematic review and meta-analysis of cohort studies using consensus definitions of exposure. Kidney Int. 2019 Jan;95(1):160-172. doi: 10.1016/j.kint.2018.08.036. Epub 2018 Nov 23. PMID 30473140